CLINICAL TRIAL: NCT01492647
Title: A Randomized, Double Blinded, Single Topical Dose Study of JNJ 10229570-AAA to Evaluate Safety and Tolerability in Japanese Subjects With Acne Vulgaris
Brief Title: A Study of JNJ 10229570-AAA to Evaluate Safety and Tolerability in Japanese Participants With Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR018673; 10229570-JPN-02 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; JNJ 10229570-AAA; Japanese patients; Topical treatment
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JNJ 10229570-AAA 1.2% (Experimental)
  Interventions: Drug: JNJ 10229570-AAA 1.2%; Drug: Color-matched vehicle containing 0 mg of JNJ 10229570-AAA
- JNJ 10229570-AAA 3.6% (Experimental)
  Interventions: Drug: JNJ 10229570-AAA 3.6%; Drug: Color-matched vehicle containing 0 mg of JNJ 10229570-AAA

INTERVENTIONS:
Drug: JNJ 10229570-AAA 1.2% — One single application of 2.5 mL of the cream will be applied to the face, neck, shoulders, chest and to the upper back areas.
  Arms: JNJ 10229570-AAA 1.2%
Drug: JNJ 10229570-AAA 3.6% — One single application of 2.5 mL of the cream will be applied to the face, neck, shoulders, chest and to the upper back areas.
  Arms: JNJ 10229570-AAA 3.6%
Drug: Color-matched vehicle containing 0 mg of JNJ 10229570-AAA — One single application of 2.5 mL of the color-matched vehicle will be applied to the face, neck, shoulders, chest and to the upper back areas.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of JNJ 10229570-AAA after a single topical application of JNJ 10229570-AAA 1.2% and 3.6% cream in Japanese participants with acne.

DETAILED DESCRIPTION:
This is a randomized (drug assigned by chance like flipping a coin), double blinded (neither physician nor patient knows the name of the assigned drug), single dose ascending study of JNJ 10229570-AAA in Japanese participants with acne. The study will evaluate the safety and pharmacokinetics ([PK] how the drug is absorbed in the body, how it is distributed within the body and removed from the body over time) of M1 (active metabolite) in a total of eighteen (18) participants enrolled in the study, nine (9) in each group. Each participant will receive JNJ 10229570-AAA at 1.2%, 3.6% or vehicle in a cream formulation as a 2.5 mL application, to the face, neck, shoulders, chest and upper back areas. The investigational product will be washed off after the blood sampling at 24 hours after application. Safety and tolerability will be evaluated throughout the study and a topical dermatological assessment will be done by the dermatologists. The total duration of the study will be maximum 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Have Acne vulgaris, presenting at least inflammatory lesion on the face
* Body mass index between 18.0 and 30.0 kg/m2 (inclusive), and body weight not less than 50 kg (man) or 45 kg (woman)
* Blood pressure between 90 and 140 mmHg systolic (inclusive), and no higher than 90 mmHg diastolic
* Electrocardiogram (ECG) consistent with normal cardiac conduction and function
* Non-smoker
* Adequate contraception method for both men and women. If a woman, must have a negative pregnancy test
* Signed an informed consent document

Exclusion Criteria:

* History of or current clinically significant medical illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, biochemistry or urinalysis
* Clinically significant abnormal physical examination, vital signs or ECG - Use of any prescription or nonprescription medication within 14 days before the study treatment
* History of drug or alcohol abuse within the past 5 years
* Drug allergy or drug hypersensitivity
* Blood donation, depending on the volume of blood collection
* Positive test for human immunodeficiency virus (HIV), hepatitis B or C, or syphilis
* Dermatological disease at application site
* Photosensitivity
* Exposure to excessive or chronic ultraviolet (UV) radiation (i.e., sunbathing, tanning salon use, phototherapy) within 4 weeks prior to study treatment or planned during the study period

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Topical Dermatological Assessment (Scores on Scales) | Days 1-7
  The Topical Dermatological Assessment is based on the 3 to 4-point Cutaneous Irritation Grading Scales that assess the level of Erythema, Dryness, Peeling/Scaling, Burning/Stinging, and Itching from 0 (no reaction) to 3 or 4 (strong reaction). In addition, the assessment observes and records any pigmentation change that may occur on the skin after the intervention.

SECONDARY OUTCOMES:
Plasma M1 concentrations | 12 time points up to 72 hours
PK parameters | 12 time points up to 72 hours
  PK parameters of JNJ-10229570-AAA, as measured by AUC, Cmax and tmax

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (2):
- Japan (2):
  - Fukukoka
  - Hakata